CLINICAL TRIAL: NCT00894933
Title: Performance Evaluation of the AMS CONTINUUM™ Device in Facilitating Vesico-Urethral Anastomosis Following a Radical Prostatectomy
Brief Title: Performance Evaluation of the AMS CONTINUUM™ Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PE0814; G090011
Record Dates: First submitted 2009-05-05; First posted 2009-05-07 (Estimated); Results first posted 2017-03-13 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2017-01

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Radical Prostatectomy; Vesico-Urethral Anastomosis
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Continuity of Patient Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Continuum (Experimental): Verify the consistency of performance of the AMS CONTINUUM device in facilitating a sustainable anastomosis following a radical prostatectomy using updated Device design elements and Physician training materials on Device implant technique.
  Interventions: Device: CONTINUUM™

INTERVENTIONS:
Device: CONTINUUM™ — Performance of CONTINUUM™ in facilitating the vesico-urethral anastomosis following radical prostatectomy.
  Other Names: Anastomosis Device

SUMMARY:
1. To assess the safety of using the CONTINUUM™ device by monitoring the side effects and complications associated with the Device following a radical prostatectomy.
2. To verify CONTINUUM™ device performance using updated CONTINUUM™ device design modifications, physician procedure guide and training methodology.

DETAILED DESCRIPTION:
Surgery is the main treatment for localized prostate cancer. The most common technique is a "radical prostatectomy," which involves removing the prostate gland, seminal vesicles and nearby lymph nodes. Radical prostatectomy is a major operation, most suitable for otherwise healthy men whose cancer does not appear to have spread.One of the most technically challenging aspects of this surgery is reconstruction of the interrupted urinary tract by hand suturing the bladder neck anastomosis, in which the bladder neck is sewn to the urethra after the prostate has been removed.

CONTINUUM™ (study Device) is a surgical device intended to be used as part of the radical prostatectomy procedure. The Device facilitates approximation of the bladder neck and urethral stump by bringing together and holding the tissue in place until adequate natural healing of the vesico-urethral anastomosis occurs. CONTINUUM™ also approximates the bladder and urethral stump to minimize extravasation, while simultaneously providing a conduit for drainage of urine from the bladder while the anastomotic site heals.

The concept of the CONTINUUM™ device and the feasibility of its operation have been tested in animal and human studies. Pilot clinical studies in the United States (G060095) found that the majority of Subjects who received and were discharged with the Device demonstrated a water-tight vesico-urethral anastomosis at the first Device removal visit. Additionally, no unanticipated adverse device effects (UADEs) were reported. The intent of this study is to verify CONTINUUM™ device performance across a variety of US sites and physicians using updated CONTINUUM™ device design modifications and physician training methodology on Device implant and removal techniques prior to initiation of a randomized US Pivotal study.

ELIGIBILITY:
Inclusion Criteria:

* All males ≥ 40 years old who are indicated for a radical prostatectomy will be eligible to participate in the study.
* The Subject is willing and able to return for study follow-up visits according to the protocol.
* The Subject can be off diuretics and blood thinners for at least one week prior to surgery.

Exclusion Criteria:

* If contraindicated for surgery
* Inability to understand the study or a history of non-compliance with medical advice
* Unwilling or unable to sign an Informed Consent Form (ICF)
* Participation in another clinical trial
* Previously implanted urological device
* A history of Recurrent urinary tract infections (UTI)
* A history of stricture disease
* Prior invasive prostate treatments (e.g., TURP, TUIP, laser therapy, radiotherapy, cryotherapy)
* Neurological disease with a history of bladder dysfunction (e.g., Parkinson's disease)
* Uncontrolled insulin-dependent diabetes
* Chemotherapy within the past 6 months
* Non-topical steroid use within the past 6 months
* History of connective tissue or autoimmune conditions
* Compromised immune system
* Allergy to nitinol, nickel, titanium or silicone
* Body Mass Index greater than or equal to 30
* American Society of Anesthesiologists Score of > 3
* Prostate size greater than or equal to 50 grams as determined by TRUS

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2009-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naveen Kella, MD, Principal Investigator — Urology San Antonio Research PA; John Libertino, MD, Principal Investigator — Lahey Clinic Medical Center
Locations (6):
- United States (6):
  - Arkansas Urology, Little Rock, Arkansas
  - Lahey Clinic Medical Center, Burlington, Massachusetts
  - Center for Urology, Rochester, New York
  - Urologic Consultants of Southeastern Pennsylvania, Philadelphia, Pennsylvania
  - Urology Clinics of North Texas, Dallas, Texas
  - Urology San Antonio Research PA, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Continuum
Started | 33
Completed | 29
Not Completed | 4
Not completed — Lost to Follow-up | 2
Not completed — Cancelled Procedure | 1
Not completed — Did not meeting incl/excl criteria | 1

BASELINE CHARACTERISTICS:
Population: Male patients ≥ 40 years old indicated for radical prostatectomy
Groups:
- Continuum Device: Performance evaluation of the AMS Continuum device in facilitating vesico-urethral anastomosis following a radical prostatectomy
Arm/Group | Continuum Device
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 33
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 33
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 27.3 (3.0)
History of smoking [Count of Participants; unit: Participants] | 19
Prostate size (g) via TRUS [Mean (Standard Deviation); unit: grams] | 33.7 (7.9)

OUTCOME MEASURES:

1. Primary Outcome: Safety - Infection That Requires IV Antibiotics or Re-hospitalization
Description: Safety of the device was evaluated by incidences of specific serious Device-related adverse complications that occurred during placement, wearing of the CONTINUUM device and during 6-month follow-up.
Time Frame: At Device placement, Device removal, 4 weeks post-Device removal, 6 months post-Device removal
Population: Subjects in whom device placement was attempted
Measure: Number; unit: Events
Arm/Group | Continuum Device
Number analyzed (Participants) | 31
Events | 0

2. Primary Outcome: Successful Device Placement
Description: Defined as the establishment of a water-tight anastomosis immediately post-Device placement.
Time Frame: At Device placement
Population: Subjects in whom device placement was attempted (i.e. treated subjects)
Measure: Count of Participants; unit: Participants
Arm/Group | Continuum Device
Number analyzed (Participants) | 31
Participants
  Successful | 30
  Not successful | 1

3. Primary Outcome: Functionally Adequate Vesico-urethral Anastomosis Within 21 Days Post-Device Placement in Subjects With Successful Device Placement
Description: Evaluated by the proportion of Subjects who have had a successful Device placement and developed a functionally adequate anastomosis within 21 days post procedure (i.e. minimal or no extravasation noted during post-placement)
Time Frame: 7-21 days post-Device placement
Measure: Count of Participants; unit: Participants
Arm/Group | Continuum Device
Number analyzed (Participants) | 30
Participants
  Successful removal at 21 days | 29
  Device not effective | 1

4. Secondary Outcome: Intraoperative/Postoperative Parameters - Estimated Blood Loss
Description: To assess short-term clinical outcomes of the Device in facilitating the vesico-urethral anastomosis following a radical prostatectomy such as blood loss.
Time Frame: At Device placement
Population: Subjects in whom device placement was attempted
Measure: Mean (Standard Deviation); unit: cc
Arm/Group | Continuum Device
Number analyzed (Participants) | 31
cc | 168.5 (219.6)

5. Secondary Outcome: Extravasation During Post-placement Cystogram at Either the First or Second Device Removal Attempts
Time Frame: 7-10 and 13 - 15 days post-Device placement
Population: Subjects with successful device placement
Measure: Count of Participants; unit: Participants
Arm/Group | Continuum Device
Number analyzed (Participants) | 30
Participants
  Successful removal at 7 - 10 days | 24
  Successful removal at 14 days | 3
  Successful removal at 21 day | 2
  Disrupted anastomosis requiring surgical intervent | 1

6. Secondary Outcome: Intraoperative/Postoperative Parameters - Total Device Placement Time
Description: To assess short-term clinical outcomes of the Device in facilitating the vesico-urethral anastomosis following a radical prostatectomy such as length of Device placement.
Time Frame: At Device placement
Population: Subjects in whom device placement was attempted
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Continuum Device
Number analyzed (Participants) | 31
Minutes | 7.4 (5.6)

7. Secondary Outcome: Intraoperative/Postoperative Parameters - Total Radical Prostatectomy Operative Time
Description: To assess short-term clinical outcomes of the Device in facilitating the vesico-urethral anastomosis following a radical prostatectomy such as length of RP procedure.
Time Frame: At Device placement
Population: Subjects in whom device placement was attempted
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Continuum Device
Number analyzed (Participants) | 31
Minutes | 142.8 (34.3)

8. Primary Outcome: Safety - Perforation of the Bowel or Bladder
Description: as for outcome 1
Time Frame: At Device placement, Device removal, 4 weeks post-Device removal, 6 months post-Device removal
Population: Subjects in whom device placement was attempted
Measure: Number; unit: Events
Arm/Group | Continuum Device
Number analyzed (Participants) | 31
Events | 1

9. Primary Outcome: Safety - Creation of a False Passage
Description: as for outcome 1
Time Frame: At Device placement, Device removal, 4 weeks post-Device removal, 6 months post-Device removal
Population: Subjects in whom device placement was attempted
Measure: Number; unit: Events
Arm/Group | Continuum Device
Number analyzed (Participants) | 31
Events | 1

10. Primary Outcome: Safety - Urinary Retention Requiring Catheterization Post-Device Removal
Description: as for outcome 1
Time Frame: At Device placement, Device removal, 4 weeks post-Device removal, 6 months post-Device removal
Population: Subjects in whom device placement was attempted
Measure: Number; unit: Events
Arm/Group | Continuum Device
Number analyzed (Participants) | 31
Events | 0

11. Primary Outcome: Safety - Mechanical Failure, Extrusion, Erosion, or Migration of the Device Requiring Surgical or Medical Intervention
Description: as for outcome 1
Time Frame: At Device placement, Device removal, 4 weeks post-Device removal, 6 months post-Device removal
Population: Subjects in whom device placement was attempted
Measure: Number; unit: Events
Arm/Group | Continuum Device
Number analyzed (Participants) | 31
Events | 0

12. Primary Outcome: Safety - Separation/Disruption of the Anastomosis Requiring Corrective Intervention
Description: as for outcome 1
Time Frame: At Device placement, Device removal, 4 weeks post-Device removal, 6 months post-Device removal
Population: Subjects in whom device placement was attempted
Measure: Number; unit: Events
Arm/Group | Continuum Device
Number analyzed (Participants) | 31
Events | 1

13. Primary Outcome: Safety - Bladder Neck Contracture
Description: as for outcome 1
Time Frame: At Device placement, Device removal, 4 weeks post-Device removal, 6 months post-Device removal
Population: Subjects in whom device placement was attempted
Measure: Number; unit: Events
Arm/Group | Continuum Device
Number analyzed (Participants) | 31
Events | 6

ADVERSE EVENTS:
Time Frame: Adverse events were collected that occurred during placement, wearing of the CONTINUUM device and during the 6-month follow-up
Arm/Group | Continuum Device
Serious Adverse Events (participants affected / at risk) | 3/31
Other Adverse Events (participants affected / at risk) | 30/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continuum Device (N=31)
Excessive bleeding (Surgical and medical procedures) | 2 (2)
Bladder Neck Contracture/Outlet Obstruct (Renal and urinary disorders) | 1 (1)
Separation/Disruption of Anastomosis (Renal and urinary disorders) | 1 (1)
Syncope (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continuum Device (N=31)
Urinary Incontinence - De Novo (Renal and urinary disorders) | 25 (26)
Pain/Discomfort (General disorders) | 12 (12)
Pain/Discomfort - Other (General disorders) | 10 (13)
Hematuria (Renal and urinary disorders) | 6 (8)
Erectile Dysfunction - De Novo (Reproductive system and breast disorders) | 18 (18)
Pain/Discomfort - Abdominal (Gastrointestinal disorders) | 8 (8)
Erectile Dysfunction - Worsening (Reproductive system and breast disorders) | 3 (3)
Infection (Infections and infestations) | 3 (3)
Urinary Tract Infection (UTI) (Infections and infestations) | 3 (3)
Urinary Retention (Renal and urinary disorders) | 2 (2)
Dysuria (Renal and urinary disorders) | 1 (1)
False Passage (Renal and urinary disorders) | 1 (1)
Perforation - Bladder (Renal and urinary disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Pain/Discomfort - Back (Musculoskeletal and connective tissue disorders) | 2 (2)
Nocturia (Renal and urinary disorders) | 2 (2)
Dizziness (General disorders) | 1 (2)
Abdominal Bloating/Gas (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Fluid Overload (Hypervolemia) (Vascular disorders) | 1 (1)
Loss of appetite (Gastrointestinal disorders) | 1 (1)
Actelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bladder Spasm (Renal and urinary disorders) | 1 (1)
Clot in catheter (Renal and urinary disorders) | 1 (1)
Disease progession (Renal and urinary disorders) | 1 (1)
Hemorrhoid (General disorders) | 1 (1)
Increased Creatinine (Renal and urinary disorders) | 1 (1)
Inguinal Hernia (Musculoskeletal and connective tissue disorders) | 1 (1)
Kidney Stone (Renal and urinary disorders) | 1 (1)
Light Headed (General disorders) | 1 (1)
Tunnel Vision (Eye disorders) | 1 (1)
Vasovagal Reaction (Cardiac disorders) | 1 (1)
Bladder Neck Contracture/Outlet Obstruct (Renal and urinary disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No